CLINICAL TRIAL: NCT02854943
Title: The Prognostic and Diagnostic Value of Ferritin in Critically Ill Patients With Special Focus on Underlying Hemophagocytic Lymphohistiocytosis
Brief Title: Investigation of Ferritin in Critically Ill Patients With Hemophagocytic Lymphohistiocytosis
Acronym: FERRITS
Status: Completed | Type: Observational
Sponsor: Gunnar Lachmann (Other)
Responsible Party: Sponsor-Investigator, Gunnar Lachmann, Specialist in Anesthesiology of the Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: HLH
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Hemophagocytic Lymphohistiocytosis (HLH); Macrophage Activation Syndrome (MAS); Hemophagocytic Syndromes
Keywords: Ferritin; Hemophagocytic lymphohistiocytosis (HLH); Critically ill patients; intensive care unit (ICU); Outcome; Diagnosis
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Macrophage Activation Syndrome; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critically ill patients: Male and female critically ill patients admitted to the Charité - University Medicine Berlin during 2000 and 2018.

SUMMARY:
Retrospective analysis of ferritin, outcome and HLH-criteria in critically ill patients.

DETAILED DESCRIPTION:
The study is a retrospective register study of critically ill patients from Charité - Universitätsmedizin Berlin during 2000 and 2016 that had at least one measurement of plasma ferritin. Outcome, underlying diagnoses and HLH-2004 criteria (Henter JI et al. 2007) will be analyzed and the HScore of these patients will be calculated (Fardet L et al. 2014). All recorded data of the specific admission term in ICU will be used for the analysis. No follow-up of the patients after discharge will be performed in this study. The study does not involve any randomization or any drug testing.

Update 2019: We expanded our database for the years until 2018 and also for the surgical and medical ICUs of the Charité - Universitätsmedizin Berlin (from 256 to 2623 patients).

Update 2022: A systematic literature search will be performed to find suitable validation cohorts for multicenter validation of optimized HLH diagnostic criteria, which are calculated based on our data (new secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* male and female patients
* at least one measurement of plasma ferritin

Exclusion Criteria:

-age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female critically ill patients admitted to the Charité - Universitätsmedizin Berlin during 2000 and 2018
Sampling Method: Probability Sample
Enrollment: 2623 (Actual)
Dates: Start 2000-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Mortality | Participants will be followed up for the duration of hospital stay, an expected average of two months
  A retrospective analysis of patients with available charts to determine the outcome whether patients survived the ICU or died.
Probability of having undiagnosed Hemophagocytic lymphohistiocytosis (HLH) | The participants will be followed up for the duration of hospital stay, an expected average of two months
  Retrospective analysis of available charts, underlying diagnoses, findings and blood values: HLH-2004 criteria (Henter JI et al. 2007) and HScore (Fardet L et al. 2014)

SECONDARY OUTCOMES:
Diagnoses | Participants will be followed up for the duration of hospital stay, an expected average of two months
  Retrospective analysis of available charts and underlying diagnoses
Intensive care unit stay | Participants will be followed up for the duration of intensive care unit stay, an expected average of one week
  Retrospective analysis of available charts and duration of ICU stay
Improving HLH diagnostic criteria including multicenter validation | Participants will be followed up for the duration of intensive care unit stay, an expected average of one week
  Sensitivity and specificity of HLH diagnostic criteria should be improved by calculating different cutoffs of HLH-2004 criteria. Combinations with highest sensitivity and specificity will be validated in published cohorts of HLH testing for sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Lachmann, MD, Study Director — Charité - Universitätsmedizin Berlin, Department of Anesthesiology and Operative Intensive Care Medicine; Gunnar Lachmann, MD, Study Chair — Charité - Universitätsmedizin Berlin, Department of Anesthesiology and Operative Intensive Care Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henter JI, Horne A, Arico M, Egeler RM, Filipovich AH, Imashuku S, Ladisch S, McClain K, Webb D, Winiarski J, Janka G. HLH-2004: Diagnostic and therapeutic guidelines for hemophagocytic lymphohistiocytosis. Pediatr Blood Cancer. 2007 Feb;48(2):124-31. doi: 10.1002/pbc.21039. PMID 16937360
- [Background] Fardet L, Galicier L, Lambotte O, Marzac C, Aumont C, Chahwan D, Coppo P, Hejblum G. Development and validation of the HScore, a score for the diagnosis of reactive hemophagocytic syndrome. Arthritis Rheumatol. 2014 Sep;66(9):2613-20. doi: 10.1002/art.38690. PMID 24782338
- [Derived] Knaak C, Schuster FS, Nyvlt P, Heeren P, Spies C, Schenk T, La Rosee P, Janka G, Brunkhorst FM, Lachmann G. Influence of transfusions, hemodialysis and extracorporeal life support on hyperferritinemia in critically ill patients. PLoS One. 2021 Jul 12;16(7):e0254345. doi: 10.1371/journal.pone.0254345. eCollection 2021. PMID 34252125
- [Derived] Knaak C, Nyvlt P, Schuster FS, Spies C, Heeren P, Schenk T, Balzer F, La Rosee P, Janka G, Brunkhorst FM, Keh D, Lachmann G. Hemophagocytic lymphohistiocytosis in critically ill patients: diagnostic reliability of HLH-2004 criteria and HScore. Crit Care. 2020 May 24;24(1):244. doi: 10.1186/s13054-020-02941-3. PMID 32448380
- [Derived] Knaak C, Schuster FS, Spies C, Vorderwulbecke G, Nyvlt P, Schenk T, Balzer F, La Rosee P, Janka G, Brunkhorst FM, Keh D, Lachmann G. Hemophagocytic Lymphohistiocytosis in Critically Ill Patients. Shock. 2020 Jun;53(6):701-709. doi: 10.1097/SHK.0000000000001454. PMID 31626037
- [Derived] Lachmann G, Spies C, Schenk T, Brunkhorst FM, Balzer F, La Rosee P. Hemophagocytic Lymphohistiocytosis: Potentially Underdiagnosed in Intensive Care Units. Shock. 2018 Aug;50(2):149-155. doi: 10.1097/SHK.0000000000001048. PMID 30010630